CLINICAL TRIAL: NCT01726140
Title: CPAP Reduces Hypoxemia After Cardiac Surgery (CRHACS Trial). A Randomized Controlled Trial
Brief Title: CPAP Reduces Hypoxemia After Cardiac Surgery
Acronym: CRHACS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reduction of interest and recruitment.
Sponsor: University of Turin, Italy (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Daniela Pasero, Principal Investigator, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRHACS CEI-457
Record Dates: First submitted 2012-11-06; First posted 2012-11-14 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Acute Respiratory Failure Requiring Reintubation
Keywords: intubation; respiratory failure; cardiac surgery
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATMENT (Experimental): Helmet CPAP
  Interventions: Procedure: Helmet CPAP
- CONTROL (Active Comparator): Venturi Mask
  Interventions: Procedure: Venturi Mask

INTERVENTIONS:
Procedure: Helmet CPAP — the patient will receive CPAP treatment, at a PEEP level of 10 cmH2O and a FiO2 adjusted to maintain SpO2>95%, for six hours. After three hours of treatment a blood gas analysis will be evaluated and the patient will proceed with the treatment for three more hours. At the end of the six hours, the patient will repeat a spontaneous breathing trial with a Venturi mask at FiO2 = 50%, for 15 minutes and than a blood gas analysis will be repeated: if the PaO2/FiO2 will be < 200 the patient will received a second treatment with CPAP; if PaO2/FiO2 will be >200, the patient will stop the treatment.
  Arms: TREATMENT
Procedure: Venturi Mask — the patient will maintain spontaneous breathing, with a system for oxygen delivery at a FiO2 adjusted to maintain SpO2>95%, for six hours. After three hours of treatment a blood gas analysis will be evaluated and the patient will proceed with the treatment for three more hours. At the end of the six hours, the patient will do a trial for 15 minutes and after that a blood gas analysis will be repeated: if the PaO2/FiO2 will be < 200 the patient will go on with the control treatment; if PaO2 /FiO2 will be >200, the patient will stop the treatment.
  Arms: CONTROL

SUMMARY:
The aim of study is to evaluate whether the application of a continuous positive airway pressure (CPAP) after extubation in patients undergoing cardiac surgery can reduce hypoxemia and re-intubation rate.

DETAILED DESCRIPTION:
We want to test the hypothesis that the application of a continuous positive airway pressure (CPAP) after extubation in patients undergoing cardiac surgery can reduce hypoxemia and re-intubation rate.

Primary end point: to reduce the rate of re-intubation.

Secondary end point: to reduce the incidence of atelectasis, pneumonia, sepsis, the mortality rate, the intensive care unit (ICU) and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery on cardiopulmonary bypass
* PaO2 /FiO2 < 200 after extubation
* extubation time < 24 h.

Exclusion Criteria:

* patients < 18 years old
* extracorporeal membrane oxygenation
* severe cardiac dysfunction (FE<25%)
* mechanical ventilation before the intervention
* severe COPD (patients on oxygen therapy, with a FEV1< 50%)
* heart or lung transplantation
* lack of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2023-07 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
rate of re-intubation | at 28 days

SECONDARY OUTCOMES:
incidence of atelectasis | at 28 days
incidence of pneumonia | at 28 days
incidence of sepsis | at 28 days
mortality rate | at 28 days
the intensive care unit length of stay | at 28 days
hospital length of stay | at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Vito Marco VM Ranieri, MD, Study Chair — University of Turin, Italy
Locations (1):
- University of Turin - Department of Anesthesia and Intensive Care Medicine, Turin, Italy

REFERENCES:
- [Derived] Pasero D, Costamagna A, Filippini C, Blangetti I, Cattaneo S, Baiocchi M, Balata A, Bottiroli M, Dambruoso P, De Paulis S, Grazioli L, Locatelli A, Lorini FL, Mascotti A, Mondino MG, Paparella D, Salvi L, Tonetti T, Tritapepe L, Ranieri VM. Continuous positive airway pressure to prevent reintubation in patients recovering from cardiac surgery: A multicentre randomised clinical trial. Eur J Anaesthesiol. 2025 Nov 1;42(11):958-965. doi: 10.1097/EJA.0000000000002229. Epub 2025 Jun 27. PMID 40574561